CLINICAL TRIAL: NCT03158389
Title: Umbrella Protocol for Phase I/IIa Trials of Molecularly Matched Targeted Therapies Plus Radiotherapy in Patients With Newly Diagnosed Glioblastoma Without MGMT Promoter Methylation: NCT Neuro Master Match - N²M² (NOA-20)
Brief Title: NCT Neuro Master Match - N²M² (NOA-20)
Acronym: N²M²
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: German Cancer Aid (Other); German Cancer Research Center (Other); National Center for Tumor Diseases, Heidelberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Wick, Coordinating Investigator, University Hospital Heidelberg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2014-0235/N2M2; 2015-002752-27 (EudraCT Number)
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Glioblastoma, Adult
Keywords: MGMT methylation; targeted therapy; umbrella protocol
MeSH Terms: conditions — Glioblastoma | interventions — APG101; alectinib; RG7388; atezolizumab; HhAntag691; temsirolimus; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Subtrial A: APG101 (Experimental): * weekly application of 800 mg i.v. for 6 months or until progression
  * in conjunction with radiotherapy (at 60 Gy in 2 Gy fractions) for the first 6 weeks
  Interventions: Drug: APG101
- Subtrial B: Alectinib (Experimental): * 600 mg orally twice daily (bid) for 6 months or until progression
  * in conjunction with radiotherapy (at 60 Gy in 2 Gy fractions) for the first 6 weeks
  Interventions: Drug: Alectinib
- Subtrial C: Idasanutlin (Experimental): * at escalating doses from 100 mg until maximum tolerated dose daily administered (orally) on five consecutive days of a 28-day cycle for 6 months or until progression
  * in conjunction with radiotherapy (at 60 Gy in 2 Gy fractions) for the first 6 weeks
  Interventions: Drug: Idasanutlin
- Subtrial D: Atezolizumab (Experimental): * application of 1200 mg i.v. every three weeks for 6 months or until progression
  * in conjunction with radiotherapy (at 60 Gy in 2 Gy fractions) for the first 6 weeks
  Interventions: Drug: Atezolizumab
- Subtrial E: Vismodegib (Experimental): * daily application of 150 mg orally for 6 months or until progression
  * in conjunction with radiotherapy (at 60 Gy in 2 Gy fractions) for the first 6 weeks
  Interventions: Drug: Vismodegib
- Subtrial F: Palbociclib (Experimental): * 75/100/125 mg orally once daily on 21/28 days
  * in conjunction with radiotherapy (at 60 Gy in 2 Gy fractions) for the first 6 weeks
  * followed by a 4 weeks break (after last dose of 2nd cycle)
  * and with maintenance therapy with palbociclib at 125 mg daily for 6 months or until progression
  Interventions: Drug: Palbociclib
- Subtrial G: Temsirolimus (Experimental): * weekly application of 25 mg i.v. for 6 months or until progression
  * in conjunction with radiotherapy (at 60 Gy in 2 Gy fractions) for the first 6 weeks
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: APG101 — weekly i.v.
  Arms: Subtrial A: APG101
Drug: Alectinib — twice daily (oral)
  Other Names: Alecensa
  Arms: Subtrial B: Alectinib
Drug: Idasanutlin — orally on 5 days of a 28 days cycle
  Arms: Subtrial C: Idasanutlin
Drug: Atezolizumab — i.v. every 3 weeks
  Arms: Subtrial D: Atezolizumab
Drug: Vismodegib — daily orally
  Other Names: Erivedge
  Arms: Subtrial E: Vismodegib
Drug: Temsirolimus — weekly i.v.
  Other Names: Troisel
  Arms: Subtrial G: Temsirolimus
Drug: Palbociclib — orally on 21 days of a 28 days cycle
  Other Names: Ibrance
  Arms: Subtrial F: Palbociclib

SUMMARY:
The objective of N²M² is the improvement of overall survival of patients with glioblastoma with an unmethylated MGMT promoter based on molecular characterization and use of targeted compounds in a modern trial design. The progression-free survival rate at six months (PFS-6) will be used to make decisions.

DETAILED DESCRIPTION:
Advances in the understanding of glioblastoma at a molecular level along with technological progress have led to the identification of key genetic alterations, not only in scientific projects but also in every-day clinical practice. These alterations increasingly refine the sub-classification of glioblastoma and the introduction of molecular markers in this classification, which ultimately may allow defining subset specific treatments.

The present umbrella concept for multiple biomarker-driven subtrials anchors at the Heidelberg-based INFORM registry trial in recurrent pediatric malignancies, where in analogy to NCT Neuro Master Match (N²M²) whole-exome, low-coverage whole-genome and transcriptome sequencing is used to identify targeted agents, single or in combinations according to a dedicated algorithm. It also shares conceptual similarities with international projects currently developed for lung and breast cancer. Finally, approaches to use molecular information in glioblastoma for the definition of a therapy at progression are also planned by the "Defeat Glioma" Consortium in the US and a group of excellence centers also in the US.

The N²M² concept excels the aforementioned initiatives in the strict focus on newly diagnosed patients, the option to cross-validate molecular biomarkers in an already analyzed contemporary cohort of glioblastoma patients analyzed in the German Consortium for Translational Cancer Research (DKTK) and the use of a parallel group treated with standard-of-care (SOC). Further restriction is made by the inclusion of patients only with a low likelihood to benefit from the SOC, temozolomide (TMZ) chemotherapy on the basis of O6-methylguanine-DNA-methyltransferase (MGMT) promoter methylation, allowing to replace TMZ with a molecularly targeted agent in combination with radiotherapy (RT) in each of the experimental subtrials. Replacing TMZ by an experimental agent in the primary chemo-radiotherapy has been done in at least four completed trials, albeit without pre-selection of a targeted therapy but the more opportunistic use of an available drug with no known MGMT interaction. Focusing on newly diagnosed patients not only harbors the greater likelihood of impact on the disease, but also allows addressing questions on acquired resistance in the more likely obtained tumor tissue at recurrence.

N²M² is formally divided into a DISCOVERY and a TREATMENT aspect. DISCOVERY starts with an (epigenomewide) Illumina methylation array and a panel sequencing followed by an appropriate and accepted standard method (Sanger Sequencing or Immunohistochemistry) within the scope of these methods for target validation prior to any suggestion for patient allocation into one of the subtrials. Suggestions for patients' allocation to one of the subtrials will be based on results of accepted standard methods. These data will be generated from formaline-fixed paraffine embedded (FFPE) tissue within in 2-3 weeks after surgery. The Heidelberg site has already established the next generation gene panel sequencing (used for target discovery in case of N²M²) and genome wide DNA methylation analyses for aiding daily routine. To meet the criteria for a safe use of these data for decision-making the orthogonal, standard methods performed in the Institute of Pathology are supplemented.

DISCOVERY also includes the use of whole exome, low-coverage whole-genome, and transcriptome sequencing, the methylome analysis, and gene expression arrays to find new, unexpected targets and get a more comprehensive view on affected pathways. Discovery is also the driving force behind the work on resistant tumors. The latter may result in individual treatment decisions at recurrence, knowing there are no relevantly active treatments in this setting.

TREATMENT is driven by a match/no match decision rendered in an algorithm that will be subject to refinement in the process of the project, both by data generated in N²M², but also external evidence; i.e. there may be some linear relations between an alteration, e.g. BRAF V600E mutation and a distinct treatment or some others, but it is expected that these linear relations will be replaced in a learning system by relations that take upstream and downstream target alterations and also parallel signaling pathways into account and may therefore already predict a certain likelihood of resistance development.

In detail, FFPE tissue (and blood) from patients diagnosed with a glioblastoma harboring an unmethylated MGMT promoter after informed consent will be subjected to a (epigenomewide) methylation array and panel sequencing as well as the appropriate methods to validate any of the trial immanent targets, if they are present, with results available within a maximum of 3 weeks postoperatively. This allows for a timely decision at the molecular Neurooncology Tumor Board and a timely initiation (within 4 to 6 weeks) of the postoperative treatment. Further examinations on fresh tumor tissue (and blood) such as whole exome, low-coverage whole genome and transcriptome sequencing as well as expression arrays will be done to enhance the scientific background on the tumor tissue. These data will not be used for decision-making, Runs already done within the INFORM project with glioblastoma samples and also dry runs (n=43) for the N²M² project support the feasibility of the timelines and principal options for discovery.

Matching will be defined as a molecular situation, which makes treatment with RT and a matching targeted drug from a prespecified warehouse separated in subtrials meaningful. Patients will be informed about the identified treatment option within the "matching" open-label, parallel group Phase I/IIa trial. As for 2 of the experimental compounds (APG101 and Atezolizumab) no specific biomarker is validated at the moment, the nonmatching patients will be equally allocated to receive either APG101, Atezolizumab or the current SOC (radiochemotherapy with TMZ, TMZ-group). Patients allocated to the TMZ-group will serve as a meaningful control group with basic efficacy parameters documented, if consent has been obtained.

The objective of N²M² is the improvement of overall survival of patients with glioblastoma with an unmethylated MGMT promoter based on molecular characterization and use of targeted compounds in a modern trial design. The progression-free survival rate at six months (PFS-6) will be used to make decisions.

Parallel and ongoing translational projects within the DKTK will examine prognostic properties of the biomarkers identified to drive therapy decisions in this trial. Trial accrual will be asymmetric into the different subtrials. It is expected that 75-100 patients will be accrued into this trial per year at about 14 sites in Germany (mainly Deutsches Konsortium für Translationale Krebsforschung, DKTK and Neuroonkologische Arbeitsgemeinschaft, NOA). Importantly, the parallel SPECTAbrain initiative of the European Organization for the Research and Treatment of Cancer (EORTC) is synergistic and not competitive to our study proposal since it is focused on the treatment at recurrence, using paraffin-embedded tissues, panels/arrays only and it would be desirable that data from these initiatives are looked at in a joined manner.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed, newly diagnosed glioblastoma (astrocytoma World Health Organization (WHO) grade IV) with unmethylated MGMT promoter determined by one of the accepted methods (qPCR, pyrosequencing, methylation array) and without mutation of the isocitrate dehydrogenase genes
* Open biopsy or resection
* Craniotomy or intracranial biopsy site must be adequately healed
* Informed consent
* Standard MRI ≤ 72 (+ 12 h) post-surgery according to the present national and international guidelines
* Availability of fresh-frozen tissue, formalin-fixed, paraffin-embedded (FFPE) tissue, and blood
* Patients eligible for RT at 60 Gy in 2 Gy fractions according to the local Standard of Care
* Age: ≥18 years
* Karnofsky performance status (KPS) ≥70%
* Life expectancy > 6 months
* All female patients with reproductive potential must have a negative pregnancy test (serum or urine) within 6 days prior to start of therapy. All female patients must be surgically sterile or must agree to use adequate contraception during the period of therapy and 6 months after the end of study treatment, or women must be postmenopausal for at least 2 years. Acceptable methods of contraception comprise barrier contraception combined with a medically accepted contraceptive method for the female patient (e.g. intra-uterine device with spermicide, hormonal contraceptive since at least 2 month). Female patients must agree not to donate lactation during treatment and until 6 months after end of treatment
* Male patients willing to use contraception (condoms with spermicidal jellies or cream) upon study entry and during the course of the study and 3 months after the end of the study, have undergone vasectomy, or are practicing total abstinence. Sperm donation is not permitted for the same time interval.

Main Exclusion Criteria:

* Abnormal (≥ Grade 2 CTCAE v5.0) laboratory values for hematology, liver or renal function.
* HIV infection or active Hepatitis B or C infection, or active infections requiring oral or intravenous antibiotics or that can cause a severe disease and pose a severe danger to lab personnel working on patients' blood or tissue (e.g. rabies).
* Prior therapy for glioma (except surgery and steroids) including but not limited to carmustine wafers and immunotherapy.
* Concurrent participation in another interventional clinical trial studying a drug or treatment regimen.
* Insufficient tumor material for molecular diagnostics
* Pregnant and lactating women
* History of hypersensitivity to any of the additives of the study drug formulations
* Co-administration of anti-cancer therapies other than those administered/allowed in this study
* Any clinically significant concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study or the absorption of oral medications or that would, in the opinion of the Principal Investigator, pose an unacceptable risk to the patient in this study
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the patient before trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
PFS-6 rate | 6 months
  defined as the proportion of patients free of progression at 6 months after study entry. PFS will be calculated from study entry until clinical or radiographic progression or death, whichever comes first.Progression will be evaluated according to Response Assessment in Neurooncology (RANO) criteria or Immunotherapy Response Assessment in Neurooncology (iRANO) criteria.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (AE) | 6 months
  Toxic effects will be graded according to CTCAE v5.0.
Overall survival (OS) | 6 months
  defined as the time from first administration of the investigational medicinal product (IMP) to time of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, Prof. Dr., Principal Investigator — University Hospital Heidelberg
Locations (13):
- Germany (13):
  - Charité Berlin, Neurosurgery, Berlin
  - Knappschaftskrankenhaus Bochum GmbH, Neurology Clinic, Bochum
  - University Hospital Bonn, Neurology Clinic, Bonn
  - University Hospital Cologne, Neurosurgery, Cologne
  - University Hospital Dresden, Neurosurgery, Dresden
  - University Hospital Essen, Neurology Clinic, Essen
  - University Hospital Frankfurt, Neurooncology, Frankfurt am Main
  - University Hospital Heidelberg, Neurology Clinic, Heidelberg
  - University Hospital Saarland, Neurosurgery, Homburg
  - University Hospital Mainz, Neurosurgery, Mainz
  - University Hospital Mannheim, Neurology Clinic, Mannheim
  - University Hospital Regensburg, Neurology Clinic, Regensburg
  - University Hospital Tuebingen, Neurooncology, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wick W, Lanz LM, Wick A, Harting I, Dettmer S, Suwala AK, Ketter R, Tabatabai G, Seliger C, Glas M, Burger MC, Timmer M, Ringel FA, Mildenberger I, Schulz-Schaeffer WJ, Winkler F, Konig L, Herold-Mende C, Eisenmenger A, Pfister SM, Renovanz M, Bendszus M, Sahm F, Platten M, Kessler T. Molecularly matched targeted therapies plus radiotherapy in glioblastoma: the phase 1/2a N2M2 umbrella trial. Nat Med. 2025 Oct;31(10):3534-3541. doi: 10.1038/s41591-025-03928-9. Epub 2025 Sep 5. PMID 40913172